CLINICAL TRIAL: NCT00004999
Title: A Randomized, Double-Blind, Placebo-Controlled Study of AG1549 in Combination With Viracept (Nelfinavir Mesylate) and Combivir (Zidovudine + Lamivudine) in Treatment-Naive HIV-Infected Patients
Brief Title: Effectiveness of a New Anti-HIV Drug (AG1549) Plus Viracept (Nelfinavir) Plus Combivir (Zidovudine/Lamivudine) in HIV-Infected Patients
Status: Suspended | Phase: Phase 2 | Type: Interventional
Sponsor: Agouron Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 286C; AG1549-504
Record Dates: First submitted 2000-03-21; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-03

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Zidovudine; HIV Protease Inhibitors; Lamivudine; Disease Progression; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load; Nelfinavir; Combivir
MeSH Terms: conditions — HIV Infections; Disease Progression | interventions — lamivudine, zidovudine drug combination; capravirine; Nelfinavir

INTERVENTIONS:
Drug: Lamivudine/Zidovudine
Drug: Capravirine
Drug: Nelfinavir mesylate

SUMMARY:
The purpose of this study is to look at the effectiveness of giving a new anti-HIV drug (AG1549) plus Viracept (nelfinavir) plus Combivir (a tablet containing zidovudine plus lamivudine) to HIV-infected patients who are not taking anti-HIV drugs.

DETAILED DESCRIPTION:
[Note: As of 2/28/2001, due to toxicity studies and concerns for safety, sites were notified that they need to discontinue patients from the capravirine/placebo arms and continue patients with their background therapies or switch patients to new therapies, as deemed appropriate by the investigators.] Patients are randomized to receive Viracept plus Combivir plus either AG1549 or placebo. Patients remain on their assigned therapy for 48 weeks with one post-therapy follow-up visit. Blood samples are taken regularly to quantify plasma HIV-1 RNA, CD4 and CD8 counts, and peripheral blood mononuclear cells (PBMC). Physical exams, safety assessments, and other tests are also done throughout the study. A blood sample is taken at baseline (pre-dose) for a pharmacokinetics assessment. On Day 8 and at the end of Weeks 4, 8, 16, 24, 36, and 48, pharmacokinetic sampling is done prior to dosing and between 2 to 4 hours post-dose.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible if they:

* Are HIV-positive.
* Are at least 18 years old.
* Have a CD4 cell count of more than 50 cells/mm3.
* Have an HIV level of more than 5000 copies/ml.

Exclusion Criteria

Patients will not be eligible if they:

* Have ever taken any of the following anti-HIV drugs: nonnucleoside reverse transcriptase inhibitors (NNRTIs), AG1549, Viracept, zidovudine, lamivudine, or Combivir. Other anti-HIV drugs are allowed only if taken for no more than 30 days with the last dose taken more than 6 months prior to study entry.
* Have taken an experimental drug within 28 days of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350
Dates: Start 1999-08

CONTACTS AND LOCATIONS:
Locations (53):
- United States (46):
  - Arizona Clinical Research Ctr Inc, Tucson, Arizona
  - Univ of Southern California, Los Angeles, California
  - Highland Gen Hosp / San Francisco Gen Hosp, Oakland, California
  - ViRx Inc, Palm Springs, California
  - Research & Treatment at the California Pacific Med Ctr, San Francisco, California
  - Harbor - UCLA Med Ctr, Torrance, California
  - IDC Research Initiative, Altamonte Springs, Florida
  - Bach and Godofsky, Bradenton, Florida
  - Community Health Care, Fort Lauderdale, Florida
  - Univ of Florida, Jacksonville, Florida
  - Univ of Miami School of Medicine, Miami, Florida
  - South Shore Hosp, Miami, Florida
  - Specialty Med Care Ctrs of South Florida Inc, Miami, Florida
  - Orange County Health Dept, Orlando, Florida
  - Larry Bush, Palm Springs, Florida
  - Infectious Diseases Associates, Sarasota, Florida
  - Infectious Disease Research Institute, Tampa, Florida
  - Treasure Coast Infectious Disease Consultants, Vero Beach, Florida
  - Polk County Health Dept, Winter Haven, Florida
  - Sky Blue, Boise, Idaho
  - Northwestern Univ Med Ctr, Chicago, Illinois
  - The CORE Ctr, Chicago, Illinois
  - Indiana Univ Infectious Disease Research Clinic, Indianapolis, Indiana
  - Univ of Iowa, Iowa City, Iowa
  - Univ of Kansas School of Medicine, Wichita, Kansas
  - University of Louisville / ID Division, Louisville, Kentucky
  - HIV Outpatient Clinics / LA State Univ Med Ctr, New Orleans, Louisiana
  - Fenway Community Health Ctr, Boston, Massachusetts
  - Hawthorne Med Associates / PAACA, New Bedford, Massachusetts
  - Kansas City AIDS Research Consortium, Kansas City, Missouri
  - Univ of Nebraska Medical Ctr, Omaha, Nebraska
  - Paul Alessi, Cherry Hill, New Jersey
  - VAMC New Jersey Healthcare System, East Orange, New Jersey
  - St Mary's Hosp Family Treatment Ctr, Hoboken, New Jersey
  - Univ of Med & Dentistry of New Jersey, Newark, New Jersey
  - Bentley-Salick Medical Practice PC, New York, New York
  - Univ of Rochester Med Ctr, Rochester, New York
  - Univ of Cincinnati / Holmes Hosp, Cincinnati, Ohio
  - Med Univ of South Carolina, Charleston, South Carolina
  - Julio Arroyo, West Columbia, South Carolina
  - Southwest Infectious Diseases Associates, Dallas, Texas
  - Univ TX Galveston Med Branch, Galveston, Texas
  - Joseph C Gathe, Houston, Texas
  - Thomas Street Clinic, Houston, Texas
  - Hampton Roads Med Specialists, Hampton, Virginia
  - Wisconsin AIDS Research Consortium, Milwaukee, Wisconsin
- Canada (4):
  - Canadian HIV Trials Network, Vancouver, British Columbia
  - QEII Health Science Centre, Halifax, Nova Scotia
  - Sunnybrook Health Science Centre, Toronto, Ontario
  - Montreal Chest Institute, Montreal, Quebec
- Immunity Care and Research Inc, Santo Domingo, Dominican Republic
- Puerto Rico (2):
  - Univ of Puerto Rico School of Med, Rio Piedras
  - Clinical Research Puerto Rico Inc, San Juan